CLINICAL TRIAL: NCT05463146
Title: Effects of Deep Breathing Excercises With and Without Progressive Muscle Relaxation Technique on Post Cesarean Section Low Back Pain, Quality of Sleep and Physical Activity.
Brief Title: Effects of Deep Breathing Excer. With & Without PMR on Post C Section LBP, QOS & PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0514
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean section; Deep breathing excercises; Low back pain; Progressive muscle relaxation; Physical activity; Quality of sleep
MeSH Terms: conditions — Low Back Pain; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep breathing excercises (Experimental): Deep breathing is known as diaphragmatic breathing, is a technique that is based on the notion that mind and body integration produces relaxation technique requires participants to contract the diaphragm, slowly inhaling and exhaling. Deep breathing appears to amplify blood oxygen levels, massages the inner organs located in or close to the abdomen, and possibly stimulates the vagus nerve
  Interventions: Other: Deep breathing excercises; Other: Deep breathing exercises +and progressive muscle relaxation techniques; Other: Deep breathing exercises
- Deep breathing excercise and progressive muscle relaxation (Experimental): PMR involves participants actively contracting muscles to create tension and progressively releasing it. This routine is repeated until participants acquire complete relaxation
  Interventions: Other: Deep breathing excercises; Other: Deep breathing exercises +and progressive muscle relaxation techniques; Other: Deep breathing exercises

INTERVENTIONS:
Other: Deep breathing excercises — Deep breathing, which is also known as diaphragmatic breathing, is a technique that is based on the notion that mind and body integration produces relaxation technique requires participants to contract the diaphragm, slowly inhaling and exhaling. Deep breathing appears to amplify blood oxygen levels, massages the inner organs located in or close to the abdomen, and possibly stimulates the vagus nerve
Other: Deep breathing exercises +and progressive muscle relaxation techniques — Begin with a deep breathing exercise. Inhale deeply through your nose, feeling your abdomen rise as you fill your body with air. Then slowly exhale out the mouth, the navel pulling in toward the spine as you expel the stale air out. Repeat 3-5 cycles
Other: Deep breathing exercises — Deep breathing, which is also known as diaphragmatic breathing, is a technique that is based on the notion that mind and body integration produces relaxation technique requires participants to contract the diaphragm, slowly inhaling and exhaling. Deep breathing appears to amplify blood oxygen levels, massages the inner organs located in or close to the abdomen, and possibly stimulates the vagus nerve

SUMMARY:
To find out the Effects of deep breathing exercises with and without Progressive Muscle Relaxation Technique on Post Cesarean Section low back Pain, Quality of Sleep and Physical Activity

ELIGIBILITY:
Inclusion Criteria:

* Females who had caesarian section
* Age 20-35 years
* No contraindications to exercise stated by an obstetrician

Exclusion Criteria:

* Females having heart disease,
* Females with Diabetes mellitus,
* Pre-eclampsia or eclampsia
* Complications during the operation
* Diseases of the nervous system, e.g. MS, stroke, Respiratory diseases, Diabetes, Cancer &rheumatic diseases

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Lowback pain | 8 weeks
  The Oswestry Disability Index also known as the Oswestry Low Back Pain Disability Questionnaire and is an extremely important tool The test is considered the 'gold standard' of low back functional outcome tools.Most commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living.
Quality of sleep | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI )is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.
Physical activity | 8 weeks
  Physical activity limitation questionnaire is used to assess the limitation of physical activities due to pain after C-section. It consists of 8 items (sitting in bed, standing up, walking, performing personal hygiene, bathing, breastfeeding, eating and using a toilet) which rated as: 0= easy performed, 1= performed with difficulties, 2= performed with assistance, and 3=can't perform. The total scores ranged from 0 to 24. The women are considered to have: 0-6= No limitation of the physical activities 7-12 = Mild limitation of the physical activities 13- 18= Moderate limitation of the physical activities 19-24 = Severe limitation of the physical activities

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam Muneeb, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No